CLINICAL TRIAL: NCT04820218
Title: An Open Label Study to Evaluate At-home Testing Refraction Results With Best Corrected Visual Acuity (BCVA) Outcomes in Adults
Brief Title: At-home Testing Refraction Results With Best Corrected Visual Acuity (BCVA) Outcomes in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EyeQue Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EYEQUE - 008
Record Dates: First submitted 2021-03-23; First posted 2021-03-29 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Visual Impairment; Myopia; Hyperopia; Astigmatism
MeSH Terms: conditions — Vision Disorders; Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: Subjects who had previously tested with an EyeQue ophthalmic refraction device and ordered try-on glasses will be asked to measure their visual acuity with and without their try-on glasses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Without Try-on glasses (Other): Subjects will be asked to measure their visual acuity without their try-on glasses
  Interventions: Device: With Try-on glasses

INTERVENTIONS:
Device: With Try-on glasses — Subjects will be asked to measure their visual acuity with their try-on glasses

SUMMARY:
This study is aimed at examining the BCVA from try-on glasses constructed from measurements from the EyeQue VisionCheck.

DETAILED DESCRIPTION:
This study is aimed at examining the BCVA from try-on glasses constructed from measurements from the EyeQue VisionCheck. The refraction measurements that users obtain from the VisionCheck are from testing at-home and without additional guidance other than that normally provided to those purchasing the device.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Ages 30+
3. Had purchased an EyeQue refraction device.
4. Obtained EGN's from the EyeQue refraction device.
5. Ordered Try-On glasses based on EyeQue EyeGlass Numbers.
6. Allow use for this study the VisionCheck refraction and try-on glasses measurements, taken prior to study participation.

Subject Exclusion Criteria, Subjects that by self-report:

1. Do not have a command of the English language.
2. Lack the ability to follow instructions.
3. Lack binocular vision.
4. Are Color-blind.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Visual Acuity with and without try-on glasses | Visit 1: Day 0
  Visual Acuity with and without try-on glasses

CONTACTS AND LOCATIONS:
Overall Officials: Noam Sapiens, PhD, Principal Investigator — EyeQue Corporation
Locations (1):
- EyeQue, Newark, California, United States

IPD SHARING:
Plan to Share IPD: No